CLINICAL TRIAL: NCT06873997
Title: Analysis of the Occurrence Time of Bone Metastasis and Disease Treatment Patterns in Patients with Breast Cancer Bone Metastasis: a Retrospective Study from China
Brief Title: Real World Study of Bone Metastases in Patients with Advanced Breast Cancer
Status: Completed | Type: Observational
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Wang Xiaojia, MD, Zhejiang Cancer Hospital
Other Study IDs: IRB-2023-692
Record Dates: First submitted 2025-02-23; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer Metastatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
By analyzing the clinical data of patients with advanced breast cancer with bone metastasis admitted to our center from January 1, 2021 to February 28, 2023, this study aims to understand the real-world clinical diagnosis and treatment of breast cancer with bone metastasis, including the epidemiology of bone metastasis, screening and diagnosis methods, selection of clinical treatment methods, and occurrence of SRE. To explore the risk factors related to bone metastasis-free survival (BMFI). In addition, we will explore the use of quantitative analysis of CT values to evaluate bone metastases of breast cancer, aiming to provide a new method for imaging quantitative efficacy evaluation of bone metastases.

DETAILED DESCRIPTION:
The specific contents of our research include the basic information of breast cancer patients with bone metastasis in the early stage, neoadjuvant therapy, surgery and postoperative pathology, and adjuvant therapy; The time and location of recurrence and metastasis, treatment plan, and information related to bone metastasis include time, location, diagnosis method, treatment, occurrence of SRE, and changes in CT values of bone lesions before and after drug treatment. The objective is to understand the risk factors of bone metastasis-free survival (BMFI) of breast cancer patients with bone metastases in the real world, provide evidence and data for clinical accurate screening, observe the CT value changes of bone lesions through imaging (CT quantitative), and explore a new method for evaluating the efficacy of bone metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18y;
2. Advanced breast cancer is clearly diagnosed;
3. Imaging or pathology confirmed at least 1 bone metastasis;
4. No history of other malignant tumors at the time of initial diagnosis;
5. The physical status score of Eastern Tumor Collaboration Group (ECOG) was ≤2 points;
6. Complete clinical and follow-up data.

Exclusion Criteria:

Exclusion is defined as meeting 1 of the following exclusion criteria:

1. Patients with other malignant tumors;
2. History of hyperthyroidism and hypothyroidism, abnormal parathyroid function;
3. History of bone metabolic diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible patients admitted to Zhejiang Cancer Hospital from January 1, 2021 to February 28, 2023 were included
Sampling Method: Non-Probability Sample
Enrollment: 737 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Bone metastasis-free interval (BMFI) of breast cancer patients with bone metastasis | From the diagnosis of breast cancer to the occurrence of bone metastasis，assessed up to 100 months
  Bone metastasis-free interval (BMFI) is the time between diagnosis of breast cancer and the onset of bone metastases

SECONDARY OUTCOMES:
Number of participants with Clinical features of bone metastasis | From the diagnosis of breast cancer to the conclusion of the study period，assessed up to 100 months
  Clinical characteristics of patients with bone metastasis include age, menstrual status, body mass index (BMI), presence or non-presence of underlying disease, tumor location, primary tumor size, number of lymph node metastases, TNM stage, pathologic type, histological classification, vascular thrombus invasion, estrogen receptor (ER) status, progesterone receptor (PR) status, and other factors. Human epidermal growth factor receptor-2 (HER-2) expression, Ki-67 level, whether chemotherapy and radiotherapy, recurrence and metastasis time, recurrence and metastasis site.
Changes of CT values of bone lesions before and after treatment with bone protective drugs | From the start of treatment with bone care drugs to 1 year
  CT value selection method: A professional physician manually selected a region of interest (ROI) for a single bone metastatic lesion, and recorded the mean value of CT value, which was expressed in Hounsfield units (HU). The ROI difference of the same bone metastasis before and after treatment was not more than ±10mm2
Patterns of bone metastasis in the center | rom the diagnosis of breast cancer to the occurrence of bone metastasis,assessed up to 100 months
  The time of bone metastasis were included
Occurrence of bone-related events | From the diagnosis of breast cancer to the occurrence of bone-related events，assessed up to 100 months.
  Skeleton-relative Events (SREs) include pathological fractures, spinal cord compression, bone surgery, and radiation therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided